CLINICAL TRIAL: NCT05277649
Title: Prevention Programme for Cervicomandibular Musculoskeletal Injuries in Wind Musicians
Brief Title: Prevention of Musculoskeletal Injuries in Musicians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Margarita Pino Juste (Other)
Responsible Party: Sponsor-Investigator, Margarita Pino Juste, University Professor, University of Vigo
Organization: University of Vigo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/522
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Cervical and Mandibular Pain and Disorders in Wind Players
Keywords: Musculoskeletal pain; Neck pain; Temporomandibular disorders; Posture; Musician
MeSH Terms: conditions — Musculoskeletal Pain; Neck Pain; Temporomandibular Joint Disorders | interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: The study consists of an experimental group, which will receive an intervention, and a control group, which will neither receive nor receive any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Performance of a warm-up and cool-down exercise programme for the cervical and mandibular region before and after instrumental practice.
  Interventions: Other: Exercise programme
- Control Group (No Intervention): Participants in the control group will not make any changes in their instrumental practice habit.
  At the end of the study, participants in the control group will be asked to perform the exercises tested in the experimental group.

INTERVENTIONS:
Other: Exercise programme — Performing a programme of warm-up and stretching exercises for the cervico-mandibular region aimed at improving mobility and muscle condition.
  Other Names: Warm-up and cool-down exercise programme
  Arms: Experimental Group

SUMMARY:
Musicians are a group with a high prevalence of musculoskeletal injuries. In particular, wind musicians, due to their playing requirements, are prone to suffer from cervical and mandibular alterations.

For this reason, a specific exercise programme has been designed with the aim of analysing its effectiveness in improving these regions.

DETAILED DESCRIPTION:
This study is a clinical trial with a control group whose participants are university music students specialising in wind instrument performance.

The intervention of the participants in the Experimental Group consists of the individual performance of a specific programme of warm-up exercises prior to instrumental practice aimed at improving the mobility and strength of the cervical and mandibular regions, as well as a series of cool-down exercises after instrumental practice based on stretching the main muscles of both regions.

Participants in the Control Group will continue their normal life without performing any specific exercise previously taught by the researchers.

For the evaluation of the programme, an initial evaluation and a re-evaluation after 12 weeks will be carried out. In both, cervical and jaw mobility as well as body posture will be assessed. In addition, at the muscular level, the activity of the upper trapezius and masseter muscles will be assessed, and the pain threshold at trigger points will also be measured.

The hypotheses are that by carrying out the exercise programme designed for wind musicians, an improvement in body posture, in the range of cervical and jaw mobility and in muscle activation will be achieved, as well as a decrease in the pain threshold.

For the study of the results, an inferential statistical analysis of the data will be carried out using the Wilcoxon test for paired data or Student's t-test for repeated measures according to the sample characteristics in order to determine the effect of the exercise programme on the different variables of the experimental process. Correlation statistics will be used to establish the association between certain quantitative explanatory variables and ANOVA for categorical variables. The level of significance will be kept at p<.05 and all calculations will be carried out using the SPSS 22.0 statistical programme.

ELIGIBILITY:
Inclusion Criteria:

* Woodwind or metal musicians
* University students of music performance

Exclusion Criteria:

* Any surgical intervention in cervical spine, orofacial region or temporomandibular joint.
* Analgesics or physiotherapeutic treatment in the last 24h.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Cervical range of movement | Change from baseline at 3 months
  Evaluation of cervical range of motion (flexion-extension, tilts and rotations) with Kinovea software. The Kinovea software is a validated tool to measure the movements of the cervical spine.
Temporomandibular range of movement | Change from baseline at 3 months
  Evaluation of the maximum jaw opening with a vernier caliper. A vernier caliper is a validated tool to measure the MMO (maximum mouth opening).
Head position | Change from baseline at 3 months
  Assessment of head position by calculation of the craniovertebral angle, sagittal head angle and shoulder angle using SAPO software. SAPO is a validated tool for head posture analysis.
Head alignment | Change from baseline at 3 months
  Horizontal alignment of the head and shoulders using SAPO software. SAPO is a validated tool for head posture analysis.
Cervical and orofacial pain | Change from baseline at 3 months
  Visual Analogic Scale. The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured from 0 (no pain) to 10 (maximum pain). All the subjects will showed their pain level.

SECONDARY OUTCOMES:
Trapezius muscle activation | Change from baseline at 3 months
  EMG assessment of resting and maximal contraction activation of the trapezius muscle. Surface EMG is a validated tool for measuring muscle activation.
Masseter muscle activation | Change from baseline at 3 months
  EMG assessment of resting and maximal contraction activation of the masseter muscle. Surface EMG is a validated tool for measuring muscle activation.
Trapezius muscle pain threshold | Change from baseline at 3 months
  Pain threshold assessment at the trigger point of the upper trapezius muscle with a digital algometer. The digital algometer is a validated tool for assessing muscle pain threshold.
Masseter muscle pain threshold | Change from baseline at 3 months
  Pain threshold assessment at the trigger point of the masseter muscle with a digital algometer. The digital algometer is a validated tool for assessing muscle pain threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Pino-Juste, Professor, Study Director — University of Vigo
Locations (1):
- Facultade de Ciencias da Educación e do Deporte, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abreu-Ramos AM, Micheo WF. Lifetime prevalence of upper-body musculoskeletal problems in a professional-level symphony orchestra: Age, gender, and instrument-specific results. Medical Problems of Performing Artists. 2007; 22(3): 97-104.
- [Background] Barton R, Feinberg J. Effectiveness of an educational program in health promotion and injury prevention for freshman music majors. Medical Problems of Performing Artists. 2008; 23: 47-53.
- [Background] Elwardany SH, El-Sayed WH, Ali MF. Reliability of Kinovea Computer Program in Measuring Cervical Range of Motion in Sagittal Plane. Open Access Library Journal. 2015; 2(9): 1-10.
- [Background] García-Remeseiro T, Gutierrez-Sanchez A. Analysis of relationships between the use of visual display terminals, craniocervical angle and physical activity: A pilot study. Journal of Human Sport and Exercise. 2017; 12.
- [Background] Rodriguez-Blanco C, Cocera-Morata FM, Heredia-Rizo AM, Ricard F, Almazan-Campos G, Oliva-Pascual-Vaca A. Immediate Effects of Combining Local Techniques in the Craniomandibular Area and Hamstring Muscle Stretching in Subjects with Temporomandibular Disorders: A Randomized Controlled Study. J Altern Complement Med. 2015 Aug;21(8):451-9. doi: 10.1089/acm.2014.0332. Epub 2015 Jun 2. PMID 26218883
- [Background] Matei R, Ginsborg J. Physical Activity, Sedentary Behavior, Anxiety, and Pain Among Musicians in the United Kingdom. Front Psychol. 2020 Dec 3;11:560026. doi: 10.3389/fpsyg.2020.560026. eCollection 2020. PMID 33424675
- [Background] Ruivo RM, Carita AI, Pezarat-Correia P. The effects of training and detraining after an 8 month resistance and stretching training program on forward head and protracted shoulder postures in adolescents: Randomised controlled study. Man Ther. 2016 Feb;21:76-82. doi: 10.1016/j.math.2015.05.001. Epub 2015 May 13. PMID 26028408
- [Background] Steemers S, van Middelkoop M, de Boks GG, van Rijn RM, Bierma-Zeinstra SMA, Stubbe JH. The impact of injury definitions on measures of injury occurrence in classical music students: a prospective cohort study. BMC Musculoskelet Disord. 2020 Aug 11;21(1):534. doi: 10.1186/s12891-020-03490-0. PMID 32781988
- [Background] Steinmetz A, Moller H, Seidel W, Rigotti T. Playing-related musculoskeletal disorders in music students-associated musculoskeletal signs. Eur J Phys Rehabil Med. 2012 Dec;48(4):625-33. Epub 2012 Nov 9. PMID 23138678
- [Background] Steinmetz A, Scheffer I, Esmer E, Delank KS, Peroz I. Frequency, severity and predictors of playing-related musculoskeletal pain in professional orchestral musicians in Germany. Clin Rheumatol. 2015 May;34(5):965-73. doi: 10.1007/s10067-013-2470-5. Epub 2014 Jan 5. PMID 24389813
- [Background] Steinmetz A, Zeh A, Delank KS, Peroz I. Symptoms of craniomandibular dysfunction in professional orchestra musicians. Occup Med (Lond). 2014 Jan;64(1):17-22. doi: 10.1093/occmed/kqt148. Epub 2013 Dec 11. PMID 24336480
- [Background] van Selms MKA, Wiegers JW, van der Meer HA, Ahlberg J, Lobbezoo F, Visscher CM. Temporomandibular disorders, pain in the neck and shoulder area, and headache among musicians. J Oral Rehabil. 2020 Feb;47(2):132-142. doi: 10.1111/joor.12886. Epub 2019 Sep 24. PMID 31520546
- [Background] Zaza C, Farewell VT. Musicians' playing-related musculoskeletal disorders: an examination of risk factors. Am J Ind Med. 1997 Sep;32(3):292-300. doi: 10.1002/(sici)1097-0274(199709)32:33.0.co;2-q. PMID 9219660
- [Derived] Rodriguez-Gude C, Taboada-Iglesias Y, Pino-Juste M. Prevention of cervical and mandibular dysfunction in wind musicians: a randomized controlled trial. Int J Occup Saf Ergon. 2025 Oct 18:1-8. doi: 10.1080/10803548.2025.2564526. Online ahead of print. PMID 41108102